CLINICAL TRIAL: NCT01366040
Title: An Open-Label, Survey-Based, Multicenter Study to Determine Patient Satisfaction With Single-Use Prefilled Avonex® PEN Autoinjector in Multiple Sclerosis Patients
Brief Title: Avonex PEN Satisfaction and Patients Experience Clinical Trial
Acronym: ASPECT
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: AVX-CAN-11-08
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Sclerosis
Keywords: Patient Satisfaction; Multiple Sclerosis; Autoinjector; Avonex
MeSH Terms: conditions — Multiple Sclerosis; Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open-label, multicenter, survey-based study to determine subject satisfaction with using the single-use autoinjector for the delivery of AVONEX PS. Enrollment will consist of 200 subjects in a single cohort who have been prescribed AVONEX PEN in accord with its Product Monograph. All subjects must be experienced AVONEX PS users (i.e., using it for at least 12 weeks without any support person to help with the injections administered in the vastus lateralis) and enrolled in MS AllianceTM program (hereinafter, MS Alliance). The clinic nurse investigator will instruct the patient on the correct method of using AVONEX PEN and the first injection with Autoinjector, using the subject's own supply, will be completed in the clinic, with the clinic nurse investigator present. All further injections of AVONEX PEN will be self-administered at home. The subjects will complete the first set of questionnaires, including Subject Satisfaction Questionnaire, Ease of Use Grading Scale and the Autoinjector Instructions Grading Scale, within 10 minutes after the first injection at the clinic, and will be given another set of questionnaires to be completed at home within 10 minutes following the last study injection 2 months later, provided the subjects still continue to self-administer their AVONEX PEN. The first set of questionnaires will be left with the clinic nurse investigator to be sent to the CRO by fax or e-mail, while the second set will need to be mailed to the CRO by study subjects using the provided self-addressed, postage-paid envelope.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent. If required by local law, candidates must also authorize the release and use of Protected Health Information (PHI)
* Must be 18 to 65 years old, inclusive, at the time of informed consent
* Must be on AVONEX PS for at least 12 consecutive weeks
* Must be self-injecting AVONEX PS at the vastus lateralis site without any help, with or without use of Personal Injector
* Must be prescribed AVONEX PEN as per local labeling (Product Monograph) and enrolled in MS Alliance
* Must be able to physically demonstrate use of the Autoinjector device and be able to self-administer the injections
* Must be able to understand and comply with the protocol

Exclusion Criteria:

* Female subjects considering becoming pregnant while in the study or who are currently pregnant or breast-feeding
* Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject unsuitable for enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis (MS) subjects between the ages of 18 and 65, inclusive, who have been treated with AVONEX® PS for at least 12 weeks prior to study entry.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 2 months

SECONDARY OUTCOMES:
Ease of use grading scale | 2 months
Autoinjector instructions grading scale | 2 months

CONTACTS AND LOCATIONS:
Locations (10):
- Canada (10):
  - Foothills Medical Center, Calgary, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - MUN Hospital, Saint John's, Newfoundland and Labrador, Newfoundland and Labrador
  - Dalhousie MS Research Unit, Halifax, Nova Scotia
  - Norfolk Medical Clinic, Guelph, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique Neuro-Outaouais, Gatineau, Quebec
  - Neuro Rive-Sud, Greenfield Park, Quebec
  - IRDPQ, Québec, Quebec